CLINICAL TRIAL: NCT04515056
Title: Characterization of New Human Models of Non-histaminergic Itch and Their Interaction With the TRPM8 Receptor
Brief Title: Characterization of New Human Models of Non-histaminergic Itch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, PhD, Assistant Professor, Aalborg University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20200005
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Papain; Itch; Skin Prick Test (SPT)
MeSH Terms: conditions — Pruritus | interventions — Papain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Papain dosage (Experimental): In the 1st session, each of the middle forearms of the subject will be divided into two squared areas (4x4 cm). The two areas will be located 4 cm apart. Three areas will be exposed to 10, 50 or 100 µg of papain, while the last area will be used as control (exposed to a vehicle).
  Interventions: Drug: Papain 10 µg; Drug: Papain 50 µg; Drug: Papain 100 µg; Other: Vehicle
- Papain SPT (Experimental): Each forearm of the subject will be divided into two squared areas (4x4 cm). The provocations of three areas will be performed with 100 µg of papain by SPT lancets. To assess the potential importance of repeated pricks, papain will be applied by 1, 5 or 25 SPT pricks thought the skin. The last area will be exposed to cowage spicules (made chemically inert by autoclaving) soaked in 5 mg/ml papain solution.
  Interventions: Drug: Papain 1 SPT; Drug: Papain 5 SPT; Drug: Papain 25 SPT; Other: Cowhage

INTERVENTIONS:
Drug: Papain 10 µg — The area will be exposed to 10 µg of papain.
  Arms: Papain dosage
Drug: Papain 50 µg — The area will be exposed to 50 µg of papain.
  Arms: Papain dosage
Drug: Papain 100 µg — The area will be exposed to 100 µg of papain.
  Arms: Papain dosage
Other: Vehicle — The area will be exposed to vehicle
  Arms: Papain dosage
Drug: Papain 1 SPT — Papain will be applied by 1 SPT prick thought the skin
  Arms: Papain SPT
Drug: Papain 5 SPT — Papain will be applied by 5 SPT pricks thought the skin
  Arms: Papain SPT
Drug: Papain 25 SPT — Papain will be applied by 25 SPT pricks thought the skin
  Arms: Papain SPT
Other: Cowhage — The last area will be exposed to cowage spicules (made chemically inert by autoclaving) soaked in 5 mg/ml papain solution.
  Arms: Papain SPT

SUMMARY:
In this experiment the investigators would like to test a new new human itch model based on papain, and to characterize the sensory quality and temporary aspects of papain skin prick test (SPT) in comparison to the inactivated-cowhage delivery system.

DETAILED DESCRIPTION:
The most used model of non-histaminergic itch is cowhage but this models presents several problems, such us the impossibility of standardizing the amount of the spicules inserted in the skin and the difficulty of obtaining the substance. These aspects bring us the necessity to find a new and more standardized model of non-histaminergic itch.

Papain is a cysteine protease extracted from papaya plant that is known to cause itch if applied to the skin. For these reasons the investigators would like to test a new new human itch model based on papain, and to characterize the sensory quality and temporary aspects of papain skin prick test (SPT) in comparison to the inactivated-cowhage delivery system.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids or other addictive drugs
* Previous or current history of neurological, dermatological, immunological musculoskeletal, cardiac disorder or mental illnesses that may affect the results (e.g. neuropathy, muscular pain in the upper extremities, etc.).
* Lack of ability to cooperate
* Current use of medications that may affect the trial such as antihistamines, antipsychotics and pain killers, as well as systemic or topical steroids.
* Skin diseases
* Moles, scars or tattoos in the area to be treated or tested.
* Hypersensitivity to papaya and mango fruit, cashew nuts, rubber latex
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Superficial blood perfusion | 15 minutes
  Superficial blood perfusion is measured by a Speckle contrast imager (FLPI, Moor Instruments, England).
Measuring itch intensity by computerized Visual Analog Scale Scoring | 15 minutes
  The subjects will rate the sensation of itch on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no itch" and 100 indicates "worst itch imaginable" and similarly for sensations of stinging/pricking and burning, both of which are frequently associated with the sensation of itch.
Measuring pain intensity by computerized Visual Analog Scale Scoring | 15 minutes
  The subjects will rate the sensation of pain on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no pain" and 100 indicates "worst pain imaginable".
Measuring Alloknesis | 15 minutes
  Alloknesis is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 milliNewton of force). This stimulator is applied 0.5 cm outside the area of itch provocation.

SECONDARY OUTCOMES:
Measurement of Cold Detection Thresholds (CDT) | 15 minutes
  The tests for thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature decreases 1°C per second from a starting temperature of 32°C until the subject perceives a temperature change (cold sensation) and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 0°C will be used.
Measurement of Cold Pain Thresholds (CPT) | 15 minutes
  The tests for thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature decreases 1°C per second from a starting temperature of 32°C until the subject perceives a temperature change (cold sensation) and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 0°C will be used.
Measurement of Warm Detection Thresholds (WDT) | 15 minutes
  The tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature raises 1°C per second from a starting temperature of 32°C until the subject detects a painful sensation and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 52°C will be used.
Measurement of Heat Pain Thresholds (HPT) | 15 minutes
  The tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. During the first 8 seconds, the temperature raises 1°C per second from a starting temperature of 32°C until the subject detects a painful sensation and presses a button that will terminate the measurement and return the temperature to baseline at a rate of 5°C /s. A cut-off temperature of 52°C will be used.
Measurement of Pain to Supra-threshold Heat Stimuli | 15 minutes
  The tests will be conducted by using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. A thermode stimulator of 3x3 cm will be placed on the treated/placebo areas and kept in place by means of Velcro tape. The subjects will have to rate the pain to two suprathreshold heat pain stimuli (starting and ending at 32°C with an increase and decrease of 5°C and 3 s plateau at 50°C).
Measurement of Mechanical Pain Thresholds (MPT) | 15 minutes
  This test is conducted using a pin-prick set (Aalborg University, Aalborg).
Measurement of Mechanical Pain Sensitivity (MPS) | 15 minutes
  This test is conducted using a pin-prick set (Aalborg University, Aalborg).
Touch Pleasantness (TP) | 15 minutes
  Pleasant touch sensation measured using a standardized sensory brush (SENSELab Brush-05, Somedic AB, Hörby, Sweden) exerting a force of 200 to 400 mN.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Lo Vecchio, Principal Investigator — Aallborg University
Locations (1):
- Aalborg University, Aalborg, North Denmark, Denmark